CLINICAL TRIAL: NCT00388284
Title: Comparative Analysis of Thrombin Utilized in Endovascular Procedures of the Femoral Artery - CEASE Study
Brief Title: Safety and Efficacy Study Comparing Thrombin for Arterial Sealing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vascular Solutions LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0106
Record Dates: First submitted 2006-10-11; First posted 2006-10-16 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2008-02

CONDITIONS: Hemostasis of Arterial Punctures
Keywords: hemostasis; arterial sealing

INTERVENTIONS:
Device: Arterial Sealing

SUMMARY:
This trial is designed as a prospective, multi-center, randomized, double blinded clinical trial to evaluate the safety and efficacy of the Thrombin VSI. An immunological sub-study to assess antibody and coagulation changes in the subjects following exposure to the Vascular Solutions Diagnostic Duett Pro manufactured with Thrombin VSI and Thrombin JMI will be conducted as a component of this trial with a subset of the enrolled study subjects.

Two hundred seventy (270) subjects will be enrolled in this trial. A minimum of 50% of the subjects will be interventional subjects and up to 50% will be diagnostic subjects. All 270 subjects will provide blood specimens at baseline and at the 30 day follow-up visit for evaluation in the immunologic sub-study. Within the 270 subjects enrolled, a minimum of 45 subjects treated with the Thrombin VSI and a minimum of 45 subjects treated with the Thrombin JMI will provide blood specimens at the 60 day follow-up visit to be evaluated in the immunologic sub-study.

The primary efficacy objective is to demonstrate that the device time-to-hemostasis for the study group treated with the sealing device manufactured with Thrombin VSI is non-inferior to the study group treated with the sealing device manufactured with Thrombin JMI.

The primary safety objective is to demonstrate a device-related major complication rate for the study group treated with the sealing device manufactured with Thrombin VSI that is non-inferior to the device-related major complication rate observed for the study group treated with the sealing device manufactured with Thrombin JMI.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 years of age or older
* The subject is undergoing a diagnostic or interventional endovascular procedure via a retrograde femoral arterial access
* The subject is willing and able to provide appropriate informed consent
* The subject is willing and able to comply with the requirements of the study protocol, including the predefined follow-up evaluations

Exclusion Criteria:

Exclusion criteria determined prior to procedure:

* The subject has a history of clinically severe peripheral vascular disease documented as any of the following:

  * Severe claudication (walking < 100 feet)
  * Absent pulses in the affected limb
  * ABI < 0.5 at rest
  * Known diameter stenosis ≥ 50% in the iliac or femoral artery on the affected side
  * Prior vascular bypass surgery involving the affected femoral artery
  * Prior stent placement in the vicinity of the arterial puncture site
* The subject is known to be, or suspected to be, pregnant (verified in a manner consistent with institution's standard of care), or is lactating
* The subject has a pre-existing severe non-cardiac systemic disease or pre-existing terminal illness
* The subject has had an acute myocardial infarction ≤ 72 hours before the catheterization procedure
* The subject is unable to ambulate at baseline
* The subject is known to require an extended hospitalization (e.g., subject is undergoing CABG surgery)
* The subject has a known bleeding disorder (including thrombocytopenia [< 100,000 platelet count], thrombobasthenia, hemophilia, or von Willebrand disease)
* The subject is receiving Coumadin/warfarin therapy and has an INR > 2.0 on the day of, or the day before the study procedure. (INR of > 2.0 should not result in a dose change prior to the study procedure. If dosage changed, test should be repeated prior to the procedure)
* The subject has a known allergy to bovine derived products or any other materials used in the Diagnostic Duett Pro Sealing Device
* The subject has undergone prior use of a closure device in the ipsilateral common femoral artery ≤ 6 months before the current catheterization procedure
* The subject has undergone prior use of manual compression for closure in the ipsilateral common femoral artery ≤ 6 weeks before the current catheterization procedure
* The subject has undergone current, recent, or prior use of an intra-aortic balloon pump through the existing arterial puncture site
* The subject is unavailable for follow-up
* The subject is currently participating in another investigational device or drug trial
* The subject has previously participated in this trial (Protocol 0106)

Exclusion criteria to be determined during the procedure:

* The subject has an antegrade puncture
* The subject's arterial introducer sheath is <5F or > 9F or longer than 15.2 cm in overall length
* The subject has a suspected posterior femoral arterial wall puncture or puncture distal to the common femoral artery bifurcation
* The subject's common femoral artery diameter is estimated to be < 6 mm via angiogram
* The subject has tortuous vascular anatomy with greater than 90o bends on femoral angiogram
* The subject is severely hypertensive (defined as systolic BP > 180 mmHg or diastolic BP > 110 mmHg)
* The subject has experienced hemodynamic instability, defined as systolic blood pressure < 90 mmHg or cardiogenic shock, during or immediately post-procedure
* The subject has been anticoagulated with unfractionated heparin and has an ACT of > 300 seconds at completion of the antecedent procedure
* The subject is anticipated to continue dosing of heparin or anti-coagulant therapy (except any approved GPIIb/IIIa platelet receptor blocker) ≤ 6 hours following completion of the interventional or diagnostic procedure
* The subject has received thrombolytic therapy (e.g., streptokinase, urokinase, or t-PA) ≤ 24 hours prior to the catheterization procedure
* The subject has a large hematoma (≥ 6cm in diameter) present prior to vascular sealing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time to Hemostasis
Incidence rate of device-related major complications

SECONDARY OUTCOMES:
Time to ambulation
Subject satisfaction
Procedure success
Device success
Minor complications

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The Heart and Vascualr Institute of Florida, Safety Harbor, Florida
  - Ochsner Clinic, New Orleans, Louisiana
  - WakeMed, Raleigh, North Carolina
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Charleston Area Medica Center (CAMC), Charleston, West Virginia
  - University of Wisconsin, Madison, Wisconsin